CLINICAL TRIAL: NCT05680935
Title: The Importance of Determining the Expression Level of Various microRNAs in the Diagnosis of Atherosclerotic Plaque Instability
Brief Title: microRNAs in the Diagnosis of Atherosclerotic Plaque Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 132578
Record Dates: First submitted 2022-12-21; First posted 2023-01-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-03

CONDITIONS: Atherosclerosis of Artery
Keywords: unstable plaque; miRNA; trimethylamine N-oxide; atherosclerosis; carotid artery
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- atherosclerosis of the brachiocephalic arteries (Experimental): The recruitment of patients will be carried out at the University Clinical Hospital No. 1 of the Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University). The study will include up to 50 people - the study group with atherosclerosis of the brachiocephalic arteries.
  Interventions: Diagnostic Test: blood microRNA; Diagnostic Test: plaque and intima microRNA; Diagnostic Test: histological examination of the plaque; Diagnostic Test: blood level trimethyl N-oxide
- No brachiocephalic atherosclerosis (Experimental): The recruitment of patients will be carried out at the University Clinical Hospital No. 1 of the Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University). Up to 30 people - the control group without brachiocephalic atherosclerosis.
  Interventions: Diagnostic Test: blood microRNA; Diagnostic Test: blood level trimethyl N-oxide

INTERVENTIONS:
Diagnostic Test: blood microRNA — all patients will receive blood (20 ml) from the cubital vein for microRNA isolation.
Diagnostic Test: plaque and intima microRNA — The resulting surgical material will be sent for microRNA isolation.
  Arms: atherosclerosis of the brachiocephalic arteries
Diagnostic Test: histological examination of the plaque — The resulting surgical material (atherosclerotic plaque) will be sent for histological examination.
  Arms: atherosclerosis of the brachiocephalic arteries
Diagnostic Test: blood level trimethyl N-oxide — all patients will receive blood (20 ml) from the cubital vein for determination of plasma trimethyl N-oxide (TMAO) content.

SUMMARY:
It's a non-randomized, intervention, prospective, single-center study.

The aim of the work is to identify of biomarkers of unstable atherosclerosis in brachiocephalic arteries

Tasks:

* identify microRNAs, the expression of which is characteristic of unstable atherosclerotic lesions;
* to assess the relationship of miRNA and trimethylamine N-oxide with the progression of unstable atherosclerotic lesions;
* to determine the effect of the level of plasma trimethylamine N-oxide on the progression of atherosclerotic lesions.

DETAILED DESCRIPTION:
The recruitment of patients will be carried out at the University Clinical Hospital No. 1 of Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University). The study will include up to 50 people - the study group with atherosclerosis of the brachiocephalic arteries and up to 30 people - the control group without brachiocephalic atherosclerosis.

As part of the standard of medical care, the patient has already undergone and received the results of the following examinations before being included in the study:

* general clinical laboratory tests (complete blood count, urinalysis, low density lipoproteins, very low density lipoproteins, high density lipoproteins, total cholesterol, triglycerides, total protein, alanine aminotransferase, aspartate aminotransferase, creatinine, urea, glucose)
* ultrasound and/or multislice computed tomography (MSCT) of brachiocephalic arteries.

Patients with clinically significant atherosclerosis of the brachiocephalic arteries were hospitalized for an operation - carotid endarterectomy with obtaining surgical material (atherosclerotic plaque with adjacent intima).

Specific methods of the planned study (procedures for examination and treatment of the patient):

1. In addition, all patients will take blood (20 ml) from the cubital vein to isolate microRNAs and determine the plasma content of trimethylamine N-oxide (TMAO). The resulting surgical material will be sent for histological examination and microRNA isolation.
2. The following statistical data processing methods will be used: frequency distribution, arithmetic mean, mode, median, standard deviation, determination of normal distribution, Student's t-test, Pearson's test, Fisher's test, Spearman's correlation coefficient, multiple linear regression.

During the operation according to the standard protocol of carotid endarterectomy, an atherosclerotic plaque with a small area of adjacent intima is removed. An atherosclerotic plaque obtained during a carotid endarterectomy will be sent for histological examination to determine signs of instability. The obtained data will be compared with the level of isolated microRNAs in blood and tissue (atherosclerotic plaque, intima) to detect microRNAs, which are determined during an unstable course of the atherosclerotic process.

The data obtained will make it possible to predict the unstable course of atherosclerosis using non-invasive studies. This will allow timely detection of unstable plaques and help to make a decision and determine the tactics of managing patients with borderline sizes of atherosclerotic lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of written informed consent to participate in research work;
2. Age from 18 to 85 years;
3. Availability of data from a general blood test, blood lipid profile (total cholesterol, very low density lipoproteins, low density lipoproteins, high density lipoproteins, triglycerides);
4. Absence of clinical signs of atherosclerosis of brachiocephalic arteries (no stroke, transient ischemic attack. On auscultation of the carotid arteries, there are no additional noises);
5. Absence of signs of atherosclerosis of the brachiocephalic arteries according to ultrasound duplex scanning (USDS) and/or multispiral computed tomography (MSCT) angiography of the brachiocephalic arteries;
6. Conducted outpatient visit at a research center with clinical and biochemical blood tests performed, ultrasound examination of arterial vessels and/or multispiral tomography of arterial vessels with contrast enhancement and/or hospitalization at a research center.

Non-inclusion criteria:

1. Chronic kidney disease stage 3b and above (glomerular filtration rate < 45 ml / min / 1.73 sq.m);
2. The presence of severe somatic pathology (with the exception of atherosclerosis of the carotid arteries and conditions caused by it), reducing life expectancy to less than 6 months;
3. Chronic somatic diseases in the acute stage;
4. Weight less than 40kg and more than 125kg;
5. Pregnancy.

Exclusion Criteria

1. Refusal to continue participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
blood microRNA | at study entry, before carotid endarterectomy.
  * blood sampling from the cubital vein 20.0 ml before surgery
  * centrifuge ethylenediaminetetraacetic acid (EDTA) tubes with blood (ELMI centrifuge, Centrifuge model CM-6M) once at 1000 g for 10 minutes to sediment the cells;
  * select from above ¾ of the plasma volume, so as not to capture cells, into a new empty tube;
  * centrifuge the plasma at 2500 g for 15 minutes to sediment platelets. Remove ¾ of the supernatant without touching the pellet and transfer to a new tube. Repeat the procedure again;
  * Aliquot the supernatant taken a second time into 1.0 ml Eppendorf tubes.
  * Freeze (Thermo Scientific refrigerator-freezer) and store at -70˚C, -80˚C.
plaque microRNA | immediately after carotid endarterectomy
  - after receiving an atherosclerotic plaque and adjacent intima during the operation of carotid endarterectomy The atherosclerotic plaque obtained during the surgical intervention (carotid endarterectomy) is cut in half, the adjacent part of the intima is cut off. One half of the plaque is placed in a tube with 10% neutral buffered formalin solution and sent for histological examination. The second half and intima are placed in different test tubes with RNAprotect Tissue Reagent (Qiagen), cooled at +2 ˚С +4 ˚С, then frozen (Thermo Scientific refrigerator-freezer) and stored at -70˚С, -80˚С.
blood TMAO | at study entry, before carotid endarterectomy
  * blood sampling from the cubital vein 20.0 ml before surgery
  * centrifuge the ethylenediaminetetraacetic acid (EDTA) tube with blood (ELMI centrifuge, Centrifuge model CM-6M) at 2300 g for 15 minutes;
  * take 1.0 ml from the obtained plasma into 2 Eppendorf tubes;
  * Freeze (Thermo Scientific refrigerator-freezer) and store at -70˚C, -80˚C.
histological examination of atherosclerotic plaque | immediately after carotid endarterectomy
  - after receiving an atherosclerotic plaque and adjacent intima during the operation of carotid endarterectomy The atherosclerotic plaque obtained during the surgical intervention (carotid endarterectomy) is cut in half, the adjacent part of the intima is cut off. One half of the plaque is placed in a tube with 10% neutral buffered formalin solution and sent for histological examination.
intima microRNA | immediately after carotid endarterectomy
  * after receiving an atherosclerotic plaque and adjacent intima during the operation of carotid endarterectomy
  * the intima obtained during the surgical intervention (carotid endarterectomy) is placed in a tube with RNAprotect Tissue Reagent (Qiagen), cooled at +2 ˚С +4 ˚С, then frozen (Thermo Scientific refrigerator-freezer) and stored at -70˚С, -80˚С.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasiia Lomonosova, no, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
not recommended by the ethical committee

REFERENCES:
- See also: Multislice Computed Tomography Capabilities in Assessment of the Coronary Arteries Atherosclerotic Lesions. — http://doi.org/10.18087/cardio.2019.2.10214